CLINICAL TRIAL: NCT06299228
Title: Sensorimotor Training and Hand Therapy Versus Traditional Hand Therapy Alone Following a Distal Radius Fracture With Volar Plate Fixation: A Randomized Controlled Trial
Brief Title: Is Sensorimotor Training Effective Following a Distal Radius Fracture?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hand Surgery Associates LLC (Other)
Collaborators: Touro University Nevada (Other); Orthopaedic Specialty Group PC, Fairfield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSA
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive sensorimotor intervention and traditional hand therapy
  Interventions: Other: Experimental Group
- Control Group (Experimental): Control Group will receive Hand Therapy only
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Sensorimotor intervention, active range of motion, active assisted range of motion, strengthening
  Arms: Experimental Group
Other: Control Group — Active range of motion, active assisted range of motion and strengthening
  Arms: Control Group

SUMMARY:
The purpose of this study is to compare the short-term outcomes of individuals who have surgery (volar plate) for a wrist (distal radius) fracture who have routine hand therapy treatment versus routine hand therapy treatment and sensorimotor activities. Individuals who meet inclusion criteria at the facilities collecting data will be invited to participate. If they agree to participate, they will randomly and blindly (via concealed envelopes) be assigned to the control (routine treatment) or the sensorimotor treatment group. Data collection will occur at 3- and 6-weeks post initiation of skilled therapy and will include measurement of joint position sense, function via the Patient Rated Wrist and Hand, pain via the Numeric Pain Rating Scale, and range of motion at the digits and wrist.

DETAILED DESCRIPTION:
The study is an interventional study investigating the effectiveness of sensorimotor activities in addition to traditional occupational therapy intervention versus traditional intervention only for patients following a distal radius fracture with volar plate fixation. A convenience sample of patients from 2 outpatient orthopedic hand therapy departments will be invited to participate in the study.

The treatment for both groups will be identical with one group receiving the addition of sensorimotor activities. Participants will be divided into one of the two groups. They will be made aware that at any point they can choose to no longer participate in the study, and it will not affect their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture with volar plate fixation
* Understand English
* 18 years or older
* Available to attend skilled occupational therapy visits a minimum of 1x per week.

Exclusion Criteria:

* Prior surgery to the involved wrist/hand
* Cognitive impairment
* Distal radius fracture managed by casting or by another means of fixation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Active Joint Position Sense (AJPS) | Baseline, 3 and 6 weeks
  Range of motion measurement for the wrist, the measurements are recorded in degress of motion and the greater the number of degrees is reflective of greater sensorimotor deficit

SECONDARY OUTCOMES:
Patient Rated Wrist and Hand Evaluation | Baseline, 3 and 6 weeks
  Patient reported outcome measurement with a 0-100 range, 0 indicating no functional deficit and 100 indicating the worst functional scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hand Surgery Associates, Olyphant, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Only the researchers identified will have access to the participant data. 2 of the 3 researchers identified will be collecting the data.